CLINICAL TRIAL: NCT03255980
Title: Monocenter, Open Label Clinical Investigation on the Treatment With Xonrid®, a Medical Device for the Prevention and Treatment of Radiotherapy-induced Dermatitis, in Breast and Head & Neck Cancer Patients Receiving Curative Treatment.
Brief Title: Monocenter, Open Label Clinical Investigation on the Treatment of Radiation Induced Dermatitis With Xonrid®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HD01-16-30
Record Dates: First submitted 2017-07-06; First posted 2017-08-21 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-01

CONDITIONS: Radiodermatitis; Quality of Life
MeSH Terms: conditions — Radiodermatitis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: MONOCENTER, OPEN LABEL CLINICAL INVESTIGATION
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xonrid® (Experimental): Xonrid® is a medical device for radiation dermatitis
  Interventions: Device: Xonrid® gel; Other: Standard of Care
- Standard of Care (Active Comparator): Standard of care suggested by MASCC guidelines
  Interventions: Device: Xonrid® gel

INTERVENTIONS:
Device: Xonrid® gel — Water based gel for the management of toxicity skin symptoms induced by Radiotherapy
Other: Standard of Care — Standard of care suggested by MASCC' Skyn Toxicity Study Group guidelines
  Arms: Xonrid®

SUMMARY:
To evaluate the performance of Xonrid® in the prevention and treatment of G2 radiation dermatitis in breast and head & neck cancer patients.

DETAILED DESCRIPTION:
The aim of this clinical investigation is to evaluate if the use of Xonrid® in the prevention and treatment of G2 radiation dermatitis in breast and head & neck cancer patients can be a valid support, when compared to the Standard of Care as defined by MASCC (Multinational Association for Supportive Care in Cancer) guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female which are 18 years of age or older
2. Performance status < 2
3. Epithelial carcinoma of oropharynx, nasopharynx, larynx, hypopharynx, paranasal sinus and salivary glands or breast cancer, planned to receive a total dose of at least 50 Gy
4. Postoperative or curative radiation treatment
5. Concurrent chemotherapy is accepted, in head & neck cancer patients
6. Patients willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the Clinical Investigation Plan tests and procedures.

Exclusion Criteria:

1. Pregnant or lactating women
2. Planned to receive concurrent cetuximab
3. Previous radiation therapy on the head and neck area or breast and thorax areas
4. Cutaneous and connective diseases (i.e. lupus erythematosus or scleroderma)
5. Systemic diseases known to delay the skin healing process such as diabetes mellitus or severe renal failure
6. Use of a tissue-equivalent bolus
7. Use of over-the-counter topical medications containing steroids
8. Presence of rashes or unhealed wounds in the radiation field
9. Recent sun exposure
10. Mental conditions that could adversely affect patients' adherence to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orlandi Ester, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FPI: June 2017 LPO: July 2018
Groups:
- Breast Cancer Group: Xonrid+SOC: Patients treated with the device under evaluation and according to MASCC guidelines
- Breast Cancer Group: SOC: Patients treated with Standard of Care according to MASCC guidelines
- Head and Neck Cancer Group: Xonrid + SOC: H&N Patients treated with the device under evaluation and according to MASCC guidelines
- Head and Neck Cancer Group: SOC: H&N Cancer Patients treated with Standard of Care according to MASCC guidelines
Period: Overall Study
Arm/Group | Breast Cancer Group: Xonrid+SOC | Breast Cancer Group: SOC | Head and Neck Cancer Group: Xonrid + SOC | Head and Neck Cancer Group: SOC
Started | 20 | 20 | 20 | 20
Completed | 17 | 12 | 14 | 8
Not Completed | 3 | 8 | 6 | 12
Not completed — Grade =>3 Skin Toxicity | 1 | 4 | 6 | 5
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Lack of compliance to study or assessmen | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Descriptive statistics of all relevant variables were performed
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Cancer Group: Xonrid+SOC | Breast Cancer Group: SOC | Head and Neck Cancer Group: Xonrid + SOC | Head and Neck Cancer Group: SOC | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.56 (4.80) | 49.01 (4.54) | 55.73 (12.46) | 59.49 (12.34) | 53.45 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 4 | 4 | 48
  Male | 0 | 0 | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: Caucasian] | 20 | 20 | 20 | 20 | 80
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Without Grade G2 Skin Toxicity Radiodermatitis at Week 5
Description: The primary endpoint of this clinical investigation was the proportion of patients without G2 radiation dermatitis (radiation dermatitis < G2) at week 5
Time Frame: 5 weeks over 7 weeks
Measure: Number; unit: participants
Groups:
- Breast Cancer Group: SOC: Patients with Breast Cancer treated with Standard of Care according to MASCC guidelines
Arm/Group | Breast Cancer Group: Xonrid+SOC | Breast Cancer Group: SOC | Head and Neck Cancer Group: Xonrid + SOC | Head and Neck Cancer Group: SOC
Number analyzed (Participants) | 18 | 18 | 20 | 16
participants | 10 | 5 | 13 | 11

2. Secondary Outcome: Median Time to G2 Radiodermatitis Development
Description: Skin toxicity assessed accoriding to CTCAE v4.0 Term Dermatitis Radiation
Time Frame: 5 weeks over 7 weeks
Reporting Status: Not Posted

3. Secondary Outcome: The Proportion of Patients Without G2 Radiation Dermatitis at Week 6 for Both Cancer Sites, at Week 7 for Head & Neck Cancer and 2 Weeks After the Last Radiation for Both Cancer Sites
Description: Definition of RD grade according to CTCAE v4.0 Scale by trained physicinans
Time Frame: 5 weeks over 7 weeks
Reporting Status: Not Posted

4. Secondary Outcome: The Worst Skin Toxicity During Treatment and Until 2 Weeks After the Last Radiation
Description: Skin toxicity assessed accoriding to CTCAE v4.0 Term Dermatitis Radiation for both cancer sites, at week 7 for head & neck cancer and 2 weeks after the last radiation for both cancer sites.
Time Frame: 6 weeks over 7 weeks
Reporting Status: Not Posted

5. Secondary Outcome: The Changes in Skin Erythema and Pigmentation, According to the ITA (Individual Typological Angle) Degrees Measured Throughout the Study.
Description: The changes in skin erythema and pigmentation, according to the ITA (individual Typological Angle) degrees measured throughout the study by the Investigators.
Time Frame: Follow-up: 2 weeks after the completion of radiation treatment
Reporting Status: Not Posted

6. Secondary Outcome: The Changes in Trans-epidermal Water Loss (TEWL) Assessed Through the Evaporation
Description: Changes of skin characteristics in terms of TEWL according to the progression of the Radiotherapy and consequent erythema
Time Frame: weekly during teratment (7 weeks)
Reporting Status: Not Posted

7. Secondary Outcome: The Mean and Worst Score of Skindex-16 Questionnaire
Description: Evaluate the patient's QoL changes occurred during the RT trough the validated self-assessed questionnaire Skindex-16
Time Frame: 5 weeks over 7 weeks
Reporting Status: Not Posted

8. Secondary Outcome: The Compliance to Experimental Treatment, Assessed Through the Number of Daily Product Applications Reported on the Patient's Diary, Compared to the Amount of Used Product
Description: Compliance is based on the total amount ( weight) of Xonrid used over the treatment period
Time Frame: 5 weeks over 7 weeks
Reporting Status: Not Posted

9. Secondary Outcome: The Patients' Global Satisfaction With Treatment, Assessed by Likert Scale
Description: Global patient's satisfaction recorded by the Linkert Scale
Time Frame: 6 weeks over 7 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 13 months
Groups:
- Breast Cancer: Xonrid® +SOC; Head and Neck Cancer: Xonrid + SOC: Xonrid® is a medical device for radiation dermatitis
  Xonrid® gel: Water based gel for the management of toxicity skin symptoms induced by Radiotherapy
  Standard of Care: Standard of care suggested by MASCC' Skyn Toxicity Study Group guidelines
- Breast Cancer: Standard Of Care; Head and Neck Cancer: Standard of Care: Standard of care suggested by MASCC guidelines
Arm/Group | Breast Cancer: Xonrid® +SOC | Breast Cancer: Standard Of Care | Head and Neck Cancer: Xonrid + SOC | Head and Neck Cancer: Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Cancer: Xonrid® +SOC (N=20) | Breast Cancer: Standard Of Care (N=20) | Head and Neck Cancer: Xonrid + SOC (N=20) | Head and Neck Cancer: Standard of Care (N=20)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hypersensitivity
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Cancer: Xonrid® +SOC (N=20) | Breast Cancer: Standard Of Care (N=20) | Head and Neck Cancer: Xonrid + SOC (N=20) | Head and Neck Cancer: Standard of Care (N=20)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Infections - pathogen unspecified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03255980/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT03255980/SAP_001.pdf